CLINICAL TRIAL: NCT01350349
Title: Home-delivered Intervention for Depressed, Cognitively Impaired Elders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01MH091045 (NIH); 1R01MH091045 (NIH)
Record Dates: First submitted 2011-05-06; First posted 2011-05-09 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Depression; Dementia; Geriatrics
Keywords: Depression; Dementia; Geriatrics
MeSH Terms: conditions — Depression; Dementia | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Problem Adaptation Therapy (PATH) (Experimental): Problem Adaptation Therapy (PATH) focuses on the subject, the caregiver, and the subject's home-environment, to encourage problem-solving and adaptive functioning. The goal of PATH is to decrease depression and disability.
  Interventions: Behavioral: Problem Adaptation Therapy (PATH)
- Supportive Therapy (Active Comparator): Supportive Therapy assists subjects in expressing their feelings and focusing on their strengths and abilities in working through current difficulties and transitions.
  Interventions: Behavioral: Supportive Therapy

INTERVENTIONS:
Behavioral: Problem Adaptation Therapy (PATH) — Problem Adaptation Therapy (PATH) focuses on the subject, the caregiver, and the subject's home-environment, to encourage problem-solving and adaptive functioning. The goal of PATH is to decrease depression and disability.
  Arms: Problem Adaptation Therapy (PATH)
Behavioral: Supportive Therapy — Supportive Therapy assists subjects in expressing their feelings and focusing on their strengths and abilities in working through current difficulties and transitions.
  Arms: Supportive Therapy

SUMMARY:
Among older adults the combination of depression, cognitive impairment (memory problems), and disability contribute to a worsening of physical and mental health and to poor treatment outcomes. Antidepressants help fewer than 40% of depressed elders with memory problems achieve remission from their depression. Interventions involving talking therapy are underdeveloped and understudied. Therefore, this research study will test the efficacy of Problem Adaptation Therapy (PATH), a new home-delivered psychosocial intervention for elders with major depression, memory problems, and disability. PATH focuses on the subject's "ecosystem" (the patient, the caregiver, and the home-environment) and targets behavioral problems related to both depression and disability.

PATH is delivered in a subject's home, where cognitively impaired, disabled elders face most of their difficulties. Local Home Delivered Meals programs will refer clients who have symptoms of depression and are interested in research. All participants will have an available caregiver (family, significant other, or professional) and will be randomized to 12 weekly sessions of PATH or Supportive Therapy, the current standard of care for talking therapy. The study will test whether home-delivered PATH is more effective than home-delivered Supportive Therapy in reducing the subjects' depression and disability and in increasing self-efficacy over the 12-week treatment period.

DETAILED DESCRIPTION:
Depression, cognitive impairment and disability often coexist in older adults and contribute to medical and psychiatric morbidity and mortality. We developed and propose to test the efficacy of a new psychosocial intervention, Problem Adaptation Therapy (PATH), for patients with major depression, cognitive impairment (up to the level of mild to moderate dementia) and disability. The proposed R01 study meets a critical need of this population, i.e. a treatment alternative for patients in whom antidepressants may have limited efficacy and for whom psychosocial interventions are underdeveloped and understudied.

The principal innovation of PATH is its personalized approach focusing on the patient's ecosystem (i.e. the patient, the caregiver, and the home-environment) and targeting behavioral problems related to both depression and disability. PATH is delivered at the patients' home, teaches the patient-caregiver dyad problem-solving skills, and incorporates environmental adaptations (including notes, signs, reminders, calendars, voice alarms) to improve the patient's functioning.

ELIGIBILITY:
Inclusion Criteria

1. Age: >64 (65 years and older).
2. Diagnosis: Major depression, unipolar as determined by the Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders (SCID), using Diagnostic and Statistical Manual for Mental Disorders (DSM)IV criteria.
3. Severity of depression: Montgomery Asberg Depression Rating Scale (MADRS) >=18.
4. Disability, i.e. impairment in at least 1 Instrumental Activity of Daily Living as measured by Philadelphia Multilevel Assessment Instrument - Instrumental Activities of Daily Living subscale (MAI-IADL).
5. Evidence of at least mild cognitive impairment but not severe impairment (Dementia Rating Scale (DRS) total score between 90 and 133 inclusive).
6. Caregiver (family member or professional) able and willing to participate in treatment.
7. Off antidepressants, cholinesterase inhibitors, or memantine or on a stable dosage for 12 weeks and no medical recommendation for change of these agents in the near future.
8. Command of English sufficient to participate in therapy and research assessments.

Exclusion Criteria

1. High suicide risk, i.e. intent or plan to attempt suicide in near future.
2. Axis I psychiatric disorder or substance abuse other than unipolar major depression, non-psychotic depression.
3. Axis II diagnosis of antisocial personality as determined by the SCID personality disorder section (using DSM-IV criteria).
4. Moderate to Severe Dementia: We will exclude participants with DRS Total Score corresponding to moderate or more severe dementia (DRS Total <=90).
5. Acute or severe medical illness (i.e., delirium, metastatic cancer, decompensated cardiac, liver or kidney failure, major surgery, stroke or myocardial infarction during the three months prior to entry); drugs known to cause depression (e.g., reserpine, alpha-methyl-dopa, steroids); or chronic addictive drug use.
6. Current involvement in psychotherapy.
7. Aphasia.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 134 (Actual)
Dates: Start 2011-04; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Depression | 12 weeks
  The primary objective is to compare the efficacy of Problem Adaptation Therapy vs. Supportive Therapy in reducing depressive symptoms over a 12-week treatment period among elders with major depression, cognitive impairment, and disability.

SECONDARY OUTCOMES:
Disability | 12 weeks
  A secondary objective is to compare the efficacy of Problem Adaptation Therapy vs. Supportive Therapy in reducing disability over a 12-week treatment period among elders with major depression, cognitive impairment, and disability.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris N. Kiosses, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Weill Cornell Medical College, New York, New York
  - Weill Cornell Medical College, White Plains, New York

IPD SHARING:
Plan to Share IPD: No